CLINICAL TRIAL: NCT01445561
Title: The Safety and the Tolerability of Ultra Low Dose Interleukin-2 in Healthy Volunteers
Brief Title: Ultra Low Dose Interleukin-2 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110268; 11-H-0268
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Hematologic Diseases
Keywords: Interleukin-2; IL-2; Stem Cells; Regulatory T Cells (T regs); Natural Killer Cells (NK cells); Healthy Volunteer; HV
MeSH Terms: conditions — Hematologic Diseases | interventions — Interleukin-2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): 100,000 international units/m2 SQ daily for 5 days
  Interventions: Drug: Interleukin-2 (100,00 IU/m(2) SQ)
- 2 (Experimental): 200,000 international units/m2 SQ daily for 5 days
  Interventions: Drug: Interleukin-2 (100,00 IU/m(2) SQ)

INTERVENTIONS:
Drug: Interleukin-2 (100,00 IU/m(2) SQ) — 100,000 International Units/m2 SQ daily for 5 days

SUMMARY:
Background:

- Interleukin-2 is a drug that can help stimulate the body s response to inflammation. High dose interleukin-2 has been used to treat different types of cancer and immune system disorders. However, it can cause frequent and often serious side effects at the doses currently used for treatment. Very low dose interleukin-2 (700 folds less than regular dose) was previously tested in cancer patients and stem cell transplant recipients. The study observed important immune changes and minimal side effects in those patients. Researchers want to test the healthy immune system's responses to very low doses of interleukin-2 to better understand how the drug works.

Objectives:

- To study the effects of very low doses of interleukin-2 on healthy volunteers.

Eligibility:

- Healthy volunteers at least 18 years of age.

Design:

* Participants will be screened with a medical history and physical exam. They will also have blood and urine samples.
* Participants will receive one of two possible very low doses of interleukin-2 every day for 5 days.
* Blood samples will be taken twice before the first dose, 1 day after the first dose, and before the next three doses. Followup blood samples will be taken on Days 7, 14, and 28 after the first dose.

DETAILED DESCRIPTION:
Interleukin 2 (IL-2, aldesleukin) was discovered as a T cell growth factor more than 30 years ago. IL-2 was the first human cytokine used therapeutically. IL-2 induces antigen specific T cells, and two important lymphocyte subsets: regulatory T cells (T-regs) and natural killer cells (NK) cells. T-regs have a critical role in self-tolerance and pathogenesis of autoimmune disease or graft versus host disease (GVHD), and they have been extensively studied in solid tumors, hematologic malignancies, viral hepatitis, and HIV infections. NK cells have a unique role in bridging innate and adaptive immunity. NK cells facilitate hematopoietic stem cell (HSC) engraftment reduce GVHD and increase graft-versus-leukemia (GVL) effects. NK cells have important roles on pathogenesis of malignancies, autoimmune disease and AIDS. Conventional dose IL-2 treatment promotes marked expansion of regulatory T cells, and NK cells but is associated with significant side effects. However, much lower doses of interleukin-2 (0.5- 1MIU/m2/day) which lack significant side effects, also induce expansion of T regs and NK cells. These observations suggest that ultra low dose IL-2 would be safe and appropriate to give to hematopoietic stem cell donors. The quality of the transplant would be improved because the higher dose of T-regs would reduce the risk of GVHD while the higher NK cells would augment the GVL effect. The aim of this study is to evaluate the safety and the tolerability of ultra low dose IL-2 in healthy volunteer for preferential expansion of T-regs and NK cells with a view to extending ultra low dose IL-2 administration to stem cell donors. We anticipate that this study will provide valuable information on the biology of IL-2 on the human immunome applicable to various human disease conditions, including cancer, immunodeficiency disease, autoimmune disease, and hematopoietic stem cell transplantation. The proposed IL-2 dose is 2-3 logs lower than the manufacturer s recommended dose. We therefore expect that the dose used in this protocol will be well tolerated. Nevertheless, because there is little information on the tolerability and safety of IL-2 at these ultra low doses, we have structured this study as a safety protocol with stopping rules for unacceptable side effects. This is important because we hope to use the safety data generated to justify a future protocol giving ultra low dose IL-2 to stem cell donors.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy volunteers confirmed by brief history and physical examination and blood work through the CHI screening protocol
* Males or females ages 18 years or older

EXCLUSION CRITERIA:

* History of inflammatory or autoimmune disease
* History of inflammatory or autoimmune disease in first degree relatives
* History of malignancies
* Recipients of hematopoietic stem cell transplant or solid organ transplant
* History of seizures
* Positive HIV, hepatitis B surface antigen or hepatitis C antibody
* History or clinical signs of cardiac disease including coronary artery disease, cardiac arrhythmia, congestive heart failure
* History or clinical signs of of pulmonary disease including obstructive lung disease and asthma
* Active infections requiring systemic antibiotic therapy or anti-viral therapy
* History of systemic fungal or mycobacterial infections
* Use of immune modifying medications, i.e.- non steroidal anti-inflammatory drugs (aspirin, ibuprofen, naproxen, celecoxib, ketrolac), steroid (prednisone, dexamethasone, hydrocortisone), chemotherapy (cisplatin, dacarbazine, interferon alpha, tamoxifen)
* Persons who are alcoholic or abusers of illicit drugs
* Female subjects who are or may be pregnant or lactating
* Psychiatric diagnoses or symptoms, to include hypomania, bipolar disorder, major depression, or dysthymia
* Abnormal or marginal peripheral blood count that in the opinion of the PI will cause Hemoglobin and Hematocrit levels to drop as a result of participation in this study
* Liver function tests above the normal laboratory reference range
* Renal function test above the normal laboratory reference range
* Contraindication to interleukin-2 (i.e. hypersensitivity to IL- 2 products, active coronary artery disease, patients with organ allograft)
* Recent recipient of any type of vaccination (i.e. rotavirus vaccine, BCG, influenza virus vaccine, rubella virus vaccine, mumps virus vaccine, measles vaccine, poliovirus vaccine, smallpox vaccine, typhoid vaccine, varicella virus vaccine, yellow fever vaccine) in the 4 weeks preceding and during active study participation
* Body mass index greater than 35
* Inability to comprehend the investigational nature of the study or provide informed consent
* Diabetes mellitus or fasting blood glucose of > 100 mg/dL.
* Any drugs or supplements that interfere with blood clotting such as Vit.E, NSAIDS, Warfarin (Coumadin), ticlopidine (Ticlid), clopidogrel (Plavix)
* Use of iodinated contrast media in the 4 weeks preceding and during active study participation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-09-28 (Actual); Primary Completion 2013-07-15 (Actual); Study Completion 2013-07-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ultra low dose IL-2. TRSAE rate of no more than 5% would allow us to proceed with future studies. | 28 days
  To determine the safety and the tolerability of ultra low dose (physiologic dose) interleukin-2 in healthy volunteers

SECONDARY OUTCOMES:
Human immune response (immunome) to ultra low dose IL-2 based on research lab assessments | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Chen Zhao, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Smith KA. Interleukin-2: inception, impact, and implications. Science. 1988 May 27;240(4856):1169-76. doi: 10.1126/science.3131876.
- [Background] Morgan DA, Ruscetti FW, Gallo R. Selective in vitro growth of T lymphocytes from normal human bone marrows. Science. 1976 Sep 10;193(4257):1007-8. doi: 10.1126/science.181845.
- [Background] Macdonald D, Jiang YZ, Gordon AA, Mahendra P, Oskam R, Palmer PA, Franks CR, Barrett AJ. Recombinant interleukin 2 for acute myeloid leukaemia in first complete remission: a pilot study. Leuk Res. 1990;14(11-12):967-73. doi: 10.1016/0145-2126(90)90109-m. PMID 2280612
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-H-0268.html